CLINICAL TRIAL: NCT05227833
Title: Vonoprazan Vs. Pantoprazole in the Prevention of Post Endoscopic Band Ligation Ulcer/Bleeding in Portal Hypertensive Patients: a Randomized Controlled Trial
Brief Title: Vonoprazan Efficacy to Prevent Post Variceal Band Ligation Ulcer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alexandria University (Other)
Collaborators: Alexandria University Hospital, Alexandria, Alexandria Governorate, Egypt (Unknown)
Responsible Party: Principal Investigator, Sameh A. Lashen, Associate Professor, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 0305413
Record Dates: First submitted 2022-01-26; First posted 2022-02-07 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Portal Hypertension; Variceal Hemorrhage; Ulcer Hemorrhage
Keywords: Portal Hypertension; Post-ligation ulcer; Vonoprazan; Pantoprazole; Variceal bleeding
MeSH Terms: conditions — Hypertension, Portal | interventions — 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine; Pantoprazole

STUDY DESIGN:
Intervention Model Description: The enrolled participants after having an endoscopic variceal ligation session will be randomly allocated to one of three interventions (for 14 days):
  Vonoprazan 20 mg once before breakfast OR Pantoprazole 40 mg before breakfast OR Placebo (no treatment) at a 1:1 ratio.
Who Masked: Investigator
Masking Description: single blinded design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Vonoprazan (Experimental): Vonoprazan (vonaspire 20 mg), tablets, one tablet per day before breakfast for 14 days starting from the day of band ligation.
  Interventions: Drug: Vonoprazan fumarate (Vonaspire)
- Pantoprazole (Active Comparator): Pantoprazole (Controloc 40 mg OR Antopral 40 mg OR Perloc 40 mg), tablets, one tablet per day before breakfast for 14 days, starting from the day of band ligation.
  Interventions: Drug: Pantoprazole 40mg
- Placebo (Placebo Comparator): No acid suppressive medications will be described.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Vonoprazan fumarate (Vonaspire) — Patients assigned to Vonoprazan (vonaspire) tablets will receive a daily dose of 20 mg before breakfast starting from the first day of band ligation.
  Other Names: Vonoprazan
  Arms: Vonoprazan
Drug: Pantoprazole 40mg — Patients assigned to Pantoprazole tablets (Controloc OR Antopral OR Perloc) will receive a daily dose of 40 mg before breakfast starting from the first day of band ligation.
  Other Names: Pantoprazole Sodium
  Arms: Pantoprazole
Other: Placebo — No Intervention
  Arms: Placebo

SUMMARY:
Endoscopic variceal ligation (EVL) is used to control and prevent variceal bleeding in patients with liver cirrhosis, but it can be complicated by bleeding from post-EVL ulcers. the current study aims at evaluating the potential benefit of different acid-suppressive therapies in prevention of post band ligation ulcer/bleeding. We will include 234 patients with cirrhotic portal hypertension undergoing endoscopic band ligation. Patients will be randomly allocated into one group of acid suppressive therapy (Vonoprazan or pantoprazole) versus placebo for 14 days. Re-endoscopy will be done after 2 weeks of treatment to assess the healing of post ligation ulcers. Any form of upper gastrointestinal bleeding will be documented.

DETAILED DESCRIPTION:
Patients with portal hypertension who have esophageal varices usually are treated by endoscopic band ligation according to the international guidelines to prevent variceal bleeding. After band ligation, patients may suffer from post-ligation ulcer and/or bleeding. In the current study, we evaluate the effectiveness of Vonoprazan, a novel potassium-competitive acid suppressor agent, in prevention of post-ligation ulcer and /or bleeding. We also will compare this drug with the proton-pump inhibitor Pantoprazole and with placebo. We aim to enroll 234 patients who will undergo elective endoscopic variceal ligation according to the BAVINO VII guidelines will be randomly assigned to one of three arms : Vonoprazan 20 mg once daily, Pantoprazole 40 mg once daily, or Placebo (no treatment). The treatment will start from the day of band ligation and will continue for 14 days. After that, a follow up endoscopy will be done to evaluate the site of band ligation. Any ulcer at the ligation site will be documented and its size will be measured. Also, any attack of bleeding from the ulcer site (if present) will be documented. A comparison between the three arms will be done in terms of effectiveness, and bleeding rates.

Safety assessment:

The safety assessment will include all patients who will receive at least 1 dose of their assigned treatment. The safety endpoints will include treatment related adverse effects (TRAEs) grouped by Medical Dictionary for Regulatory Activities version 19.1, system organ class and preferred term, and changes from baseline in an abbreviated physical examination including vital signs, signs of liver cell deterioration, and mean change in laboratory measures including hemogram, liver aminotransferases, serum urea and creatinine, liver function test.

ELIGIBILITY:
Inclusion Criteria:

* Patients with liver cirrhosis with portal hypertension who are eligible for endoscopic band ligation (Bleeding varices, or non-bleeder but with risk signs) according to BAVINO VII guidelines
* Patients who completed the study protocol.
* Eligible participants who are willing to comply with the study protocol and provide written consent.

Exclusion Criteria:

* Endoscopically confirmed pre-existing esophageal ulcers
* Ongoing therapy with any anti-acid agent,
* Hepatocellular carcinoma
* Portal vein thrombosis
* Previous anti-flux procedure,
* Barrett's esophagus,
* History of liver transplantation,
* Pregnancy, and allergy or past adverse reaction to acid-suppressive therapy
* Estimated glomerular filtration rate < 60 mL/min/1.73 meter square.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 284 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2022-11-15 (Actual)

PRIMARY OUTCOMES:
Post ligation ulcer : presence (Yes or No), number, and size | At 2 weeks after intervention (EBL)
  1. presence of post ligation ulcer (Yes/NO)
  2. the number of ulcers if present.
  3. the maximum dimension of an ulcer (if present) in millimeter.
Post endoscopic variceal ligation ulcers | At 2 weeks after intervention
  Number of participants who experienced post-ligation ulcer.
Post endoscopic variceal ligation bleeding | during the 2 weeks treatment duration
  Number of participants who experienced post-ligation ulcer bleeding.

SECONDARY OUTCOMES:
Number of participants with Vonoprazan-related adverse events as assessed by TRAEs grouped by Medical Dictionary for Regulatory Activities version 19.1 | During the 2 weeks of medication use
  * The safety assessment will include all patients who will receive at least 1 dose of their assigned treatment.
  * The safety endpoints will include treatment related adverse effects (TRAEs) grouped by Medical Dictionary for Regulatory Activities version 19.1, system organ class and preferred term, and changes from baseline in an abbreviated physical examination and laboratory parameters including:
    * Vital signs,
    * New onset hepatic encephalopathy,
    * New onset ascites OR Increasing a pre-existing ascites,
    * Changes in hemogram,
    * Liver aminotransferases,
    * Prothrombin time/INR
    * Serum Bilirubin
    * Serum urea and creatinine.
  These data will be collected through:
  * Recording the baseline clinico-laboratory parameters at the 1st visit
  * Re-evaluation of the same parameters at 2 weeks follow-up visit
  * Encouraging the patients to communication with the study team in case of any other adverse events that may occur during the treatment duration.

CONTACTS AND LOCATIONS:
Overall Officials: Sameh Lashen, MD, Principal Investigator — University of Alexandria
Locations (1):
- Alexandria Main University Hospital, Alexandria, Alexandria Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kang SH, Yim HJ, Kim SY, Suh SJ, Hyun JJ, Jung SW, Jung YK, Koo JS, Lee SW. Proton Pump Inhibitor Therapy Is Associated With Reduction of Early Bleeding Risk After Prophylactic Endoscopic Variceal Band Ligation: A Retrospective Cohort Study. Medicine (Baltimore). 2016 Feb;95(8):e2903. doi: 10.1097/MD.0000000000002903. PMID 26937932
- [Background] Lin L, Cui B, Deng Y, Jiang X, Liu W, Sun C. The Efficacy of Proton Pump Inhibitor in Cirrhotics with Variceal Bleeding: A Systemic Review and Meta-Analysis. Digestion. 2021;102(2):117-127. doi: 10.1159/000505059. Epub 2020 Feb 21. PMID 32088712